CLINICAL TRIAL: NCT06454500
Title: Randomized, Controlled Evaluations of the Effectiveness of Clinical Decision Support Systems (REEDS)
Brief Title: Clinical Decision Support to Reduce Catheter Associated Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAU3416
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Health Care Associated Infection; Catheter-associated Urinary Tract Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop Orders (Experimental): For participants in this arm, a clinical decision support tool consisting of stop orders and an expiring alert that was displayed to care team clinicians.
  Interventions: Other: Clinical decision support
- Continuous Orders (No Intervention): For participants in this arm, no clinical decision support or alerts were displayed to care team clinicians and the urinary catheter order was continuous.

INTERVENTIONS:
Other: Clinical decision support — A 48 hour expiration on orders placed for indwelling urinary catheters.
  Arms: Stop Orders

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of a clinical decision support tool consisting of a 48-hour stop order for indwelling urinary catheters versus no clinical decision support in hospitalized patients with indwelling urinary catheters. The main questions it aims to answer are:

- Does the presence of an automated stop order integrated as part of a clinical decision support tool reduce dwell time of urinary catheters and the rate of catheter associated urinary tract infections?

Participants who have indwelling urinary catheters ordered will be randomized to either have these orders automatically expire after 48 hours unless an action is taken or have orders without expiration. Researchers will compare the urinary catheter dwell time and the rate of catheter associated urinary tract infections between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital
* At least 18 years old
* Has order placed for indwelling urinary catheter

Exclusion Criteria:

* Indication for urinary catheter labeled as either "Chronic" or "Placed by urology"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79369 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Urinary catheter dwell time | Measured from time of catheter insertion until catheter removal or hospital discharge if the catheter was not removed, up to 250 days.
  The time between urinary catheter insertion and removal

SECONDARY OUTCOMES:
Catheter Associate Urinary Tract Infection (CAUTI) rate | The development of a CAUTI was assessed from time of catheter insertion until either catheter removal or hospital discharge if the catheter was not removed, up to 250 days.
  The number of CAUTI's per 1000 catheter days. CAUTIs were defined according to NHSN (National Healthcare Safety Network) criteria as a urinary tract infection where an indwelling urinary catheter (IUC) was in place for more than two consecutive days in an inpatient location on the date of event or the day before, with day of device placement being Day 1. All positive urine cultures are reviewed by members of Infection Prevention and Control to determine if they meet the defined criteria for CAUTI. Events verified as CAUTIs are then recorded in the hospital data registry. The hospital data registry was used to determine CAUTI events in this study.
CAUTI population rate | The development of a CAUTI was assessed from time of catheter insertion until either catheter removal or hospital discharge if the catheter was not removed, up to 250 days.
  The number of CAUTI's per 10000 hospital days CAUTIs were defined according to NHSN (National Healthcare Safety Network) criteria as a urinary tract infection where an indwelling urinary catheter (IUC) was in place for more than two consecutive days in an inpatient location on the date of event or the day before, with day of device placement being Day 1. All positive urine cultures are reviewed by members of Infection Prevention and Control to determine if they meet the defined criteria for CAUTI. Events verified as CAUTIs are then recorded in the hospital data registry. The hospital data registry was used to determine CAUTI events in this study.
CAUTI Free survival | The development of a CAUTI was assessed from time of catheter insertion until either catheter removal or hospital discharge if the catheter was not removed, up to 250 days.
  The time a catheter "survived" before developing a CAUTI CAUTIs were defined according to NHSN (National Healthcare Safety Network) criteria as a urinary tract infection where an indwelling urinary catheter (IUC) was in place for more than two consecutive days in an inpatient location on the date of event or the day before, with day of device placement being Day 1. All positive urine cultures are reviewed by members of Infection Prevention and Control to determine if they meet the defined criteria for CAUTI. Events verified as CAUTIs are then recorded in the hospital data registry. The hospital data registry was used to determine CAUTI events in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Adelman, MD, MS, Principal Investigator — Columbia University
Locations (8):
- United States (8):
  - NewYork-Presbyterian Westchester, Bronxville, New York
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - NewYork-Presbyterian Hudson Valley Hospital, Cortlandt Manor, New York
  - NewYork-Presbyterian Queens, Flushing, New York
  - NewYork-Presbyterian Columbia University Irving Medical Center, New York, New York
  - NewYork-Presbyterian Allen Hospital, New York, New York
  - NewYork-Presbyterian Lower Manhattan Hospital, New York, New York
  - NewYork-Presbyterian Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No